CLINICAL TRIAL: NCT05908162
Title: To Develop an Algorithm for Predicting the Unfavorable Course of Sepsis in Children Based on a Comprehensive Assessment of Immunological, Biochemical and Molecular Genetic Markers
Brief Title: Algorithm for Predicting the Unfavorable Course of Sepsis in Children
Status: Completed | Type: Observational
Sponsor: The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, E.G.Fomina, Head of the Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology
Other Study IDs: RRPCEM_SEPSIS; NCT06142162 (obsolete NCT alias)
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sepsis
Keywords: Sepsis; monocytes; neutrophils; genetic polymorphism; PDRF
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with sepsis on day 1: Patients with sepsis on day 1
  Interventions: Diagnostic Test: Bood leukocyte subsets
- Patients with sepsis on day 7: Patients with sepsis on day 7
  Interventions: Diagnostic Test: Bood leukocyte subsets
- Patients with severe bacterial infection: Patients with severe bacterial infection (pneumonia)
  Interventions: Diagnostic Test: Bood leukocyte subsets
- Patients with severe viral infection: Patients with severe viral infection (COVID19)
  Interventions: Diagnostic Test: Bood leukocyte subsets

INTERVENTIONS:
Diagnostic Test: Bood leukocyte subsets — Determination of blood leukocyte subpopulations, subpopulation of monocytes and expression CD64 on neutrophils
  Other Names: assessment of genetic polymorphism

SUMMARY:
A comprehensive strategy will be used to investigate the relationship and correlation between 4 diagnostically significant markers relevant for early diagnosis and prediction of complications and death in the development of sepsis in children (C-reactive protein, procalcitonin, presepsin and lipopolysaccharide binding protein). For the first time, an attempt will be made to assess the genetic characteristics of the patient's from the point of view of predisposition to the unfavorable development of the sepsis based on the study of polymorphism of a number of genes of the immune system (tumor necrosis factor beta; interleukin 6, 8, 10; lymphotoxin alpha, etc.).

Based on the study results, an algorithm to predict the unfavorable course of sepsis in children will be developed using a comprehensive assessment of biochemical and molecular genetic markers.

DETAILED DESCRIPTION:
* analyze biochemical markers and immune status data in sepsis patients and in the comparison group;
* assess the state of the cellular immunity, level of pro-inflammatory cytokines, genetic polymorphism of immune response genes in sepsis patients;
* carry out a correlation analysis of clinical and laboratory data and immune system among patients of different groups (with and without septic shock, taking into account the outcome);
* assess the relationship between the genetic characteristics of the patient's immune system and the severity of the pathological process;
* based on the data obtained, prepare instructions for use, which describes an algorithm to predict the unfavorable course of sepsis in children.

ELIGIBILITY:
Inclusion Criteria:

* age from 1 month to 18 years;
* confirmed septic process$
* informed consent.

Exclusion Criteria:

* age from 18 years;
* refuse of patient to participate in the trial;
* chronic mental disorders with severe manifestations;
* pregnancy/lactation;
* intercurrent severe chronic diseases;
* HIV, Hepatites B/C;
* active tuberculosis;
* cachexia of any origin;
* malignant neoplasms.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with severe viral infection, with sepsis on day 1 and day 7
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena G Fomina, Dr, Principal Investigator — The Republican Research and Practical Center for Epidemiology and Microbiology (RRPCEM)
Locations (1):
- City Children's Infectious Clinical Hospital, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Group of healthy patients
Period: Overall Study
Arm/Group | Patients With Sepsis on Day 1 | Patients With Sepsis on Day 7 | Patients With Severe Bacterial Infection | Patients With Severe Viral Infection | Control Group
Started | 50 | 47 | 33 | 20 | 35
Completed | 50 | 47 | 33 | 20 | 35
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Bood leukocyte subsets: Determination of blood leukocyte subpopulations, subpopulation of monocytes and expression CD64 on neutrophils
- Total: Total of all reporting groups
Arm/Group | Patients With Sepsis on Day 1 | Patients With Sepsis on Day 7 | Patients With Severe Bacterial Infection | Patients With Severe Viral Infection | Control Group | Total
Number analyzed (Participants) | 50 | 47 | 33 | 20 | 35 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 47 | 33 | 20 | 35 | 185
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 21 | 14 | 16 | 91
  Male | 30 | 27 | 12 | 6 | 19 | 94
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belarus | 50 | 47 | 33 | 20 | 35 | 185

OUTCOME MEASURES:

1. Primary Outcome: Blood Leukocyte Subpopulations: the Absolute Numbers of Leukocytes of Specific Phenotypes
Description: Determination of blood leukocyte subpopulations and their total number in the blood samples (10^9 cells/l): WBC (leukocytes), CD45+(lymphocytes),CD3+ (T-lymphocytes), CD3- CD16/56+ (NK-cells), CD3+ CD16/56+ (NKT-cells), CD3+ CD4+ (T-helpers), CD3+ CD8+ (T-cytotoxic cells), CD19+ (B-lymphocytes), CD14+ (monocytes): CD14+CD16- (сlassical monocytes), CD14+СD16+(Intermediate monocytes), СD14-СD16+(nonclassical monocytes).
  Leucocyte count was determined under a microscope in a Goryaev chamber.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: 10^9 cells/l
Groups:
- Patients With Sepsis, Day 1: Patients with sepsis on day 1
- Patients With Sepsis, Day 7: Patients with sepsis on day 7
Arm/Group | Patients With Sepsis, Day 1 | Patients With Sepsis, Day 7 | Patients With Severe Bacterial Infection | Patients With Severe Viral Infection | Control Group
Number analyzed (Participants) | 50 | 47 | 33 | 20 | 35
10^9 cells/l
  WBC, 10^9 cells/l | 16.0 [8.7 to 19.8] | 11.2 [7.7 to 18.6] | 11.9 [8.7 to 14.3] | 4.9 [3.8 to 7.1] | 6.9 [6.0 to 8.8]
  lymphocyte, 10^9 cells/l | 1.83 [1.23 to 3.01] | 3.10 [1.84 to 4.19] | 1.93 [0.97 to 3.02] | 1.14 [0.79 to 1.65] | 3.24 [2.44 to 3.89]
  T-lymphocytes,10^9 cells/l | 1.28 [0.65 to 2.20] | 2.0 [1.2 to 2.9] | 1.24 [0.59 to 2.32] | 0.81 [0.44 to 1.28] | 2.1 [1.64 to 2.62]
  NK-cells,10^9 cells/l | 0.10 [0.05 to 0.19] | 0.14 [0.08 to 0.35] | 0.10 [0.06 to 0.22] | 0.15 [0.09 to 0.21] | 0.36 [0.23 to 0.50]
  NKT-cells,10^9 cells/l | 0.020 [0.012 to 0.044] | 0.050 [0.026 to 0.11] | 0.025 [0.012 to 0.041] | 0.038 [0.022 to 0.071] | 0.083 [0.041 to 0.16]
  T-helpers,10^9 cells/l | 0.65 [0.34 to 1.43] | 1.0 [0.61 to 1.78] | 0.73 [0.37 to 1.68] | 0.40 [0.28 to 0.80] | 1.19 [0.89 to 1.34]
  T-cytotoxic,10^9 cells/l | 0.40 [0.21 to 0.71] | 0.69 [0.43 to 1.1] | 0.39 [0.18 to 0.66] | 0.30 [0.15 to 0.40] | 0.74 [0.55 to 0.85]
  B-lymphocytes,10^9 cells/l | 0.36 [0.17 to 0.78] | 0.54 [0.19 to 0.80] | 0.58 [0.30 to 1.0] | 0.16 [0.11 to 0.26] | 0.43 [0.24 to 0.66]
  monocytes,10^9 cells/l | 1.04 [0.35 to 1.55] | 0.78 [0.34 to 1.19] | 0.87 [0.55 to 1.50] | 0.4 [0.24 to 0.62] | 0.46 [0.35 to 0.50]
  сlassical monocytes,10^9 cells/l | 0.66 [0.27 to 1.28] | 0.45 [0.14 to 0.93] | 0.76 [0.45 to 1.26] | 0.28 [0.19 to 0.51] | 0.38 [0.28 to 0.42]
  Intermediate monocytes,10^9 cells/l | 0.09 [0.025 to 0.20] | 0.04 [0.01 to 0.09] | 0.06 [0.03 to 0.13] | 0.05 [0.03 to 0.09] | 0.027 [0.018 to 0.043]
  nonclassical monocytes,10^9 cells/l | 0.014 [0.0022 to 0.038] | 0.008 [0.001 to 0.027] | 0.015 [0.0046 to 0.048] | 0.011 [0.007 to 0.021] | 0.004 [0.003 to 0.017]
Statistical Analysis 1: Comparison: Patients With Sepsis, Day 1 vs Patients With Severe Viral Infection vs Control Group; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Blood Leukocyte Subpopulations: Flow Cytometry Measure (Percentage of Cells of Parent Population, %)
Description: Determination of the relative subpopulations of blood leukocytes (percentage of cells of parent population, %): CD45+ (% leukocytes that are lymphocytes), CD3+ (% lymphocytes that are T-cells), CD3- CD16/56+ (% lymphocytes that are NK-cells), CD3+ CD16/56+ (% T-lymphocytes that are NKT-cells), CD3+ CD4+ (% T-lymphocytes that are T-helpers), CD3+ CD8+ (% T-lymphocytes that are T-cytotoxic cells), CD19+ (% lymphocytes that are B-cells), CD14+ CD16- (% monocytes that are classical), CD14+ CD16+ (% monocytes that are intermediate), CD14- CD16+ (% monocytes that are nonclassical), nCD64+ (% neutrophils that express CD64), mHLA-DR (% monocytes that express human leukocyte antigen-DR (HLA-DR)).
  Cell samples were counted on a FACSCalibur cytofluorimeter. Data were analyzed using Flowing Software version 2.5.1 or BD FACSDiva 7.0.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: percentage of cells of parent population
Arm/Group | Patients With Sepsis, Day 1 | Patients With Sepsis, Day 7 | Patients With Severe Bacterial Infection | Patients With Severe Viral Infection | Control Group
Number analyzed (Participants) | 50 | 47 | 33 | 20 | 35
percentage of cells of parent population
  % leukocytes that are lymphocytes | 15.2 [9.9 to 25.6] | 30.3 [18.3 to 39.9] | 15.7 [11.1 to 18.9] | 24.9 [13.6 to 36.1] | 44.5 [35.4 to 52.0]
  % lymphocytes that are T-cells | 67.4 [59.1 to 77.6] | 71.5 [65.2 to 76.0] | 62.9 [57.5 to 67.9] | 69.3 [65.5 to 74.7] | 71.5 [62.9 to 76.9]
  % lymphocytes that are NK-cells | 5.42 [3.01 to 10.98] | 7.4 [4.3 to 10.2] | 4.5 [3.2 to 10.7] | 13.35 [8.79 to 18.32] | 11.6 [8.0 to 17.1]
  % T-lymphocytes that are NKT-cells | 1.19 [0.6 to 2.3] | 2.2 [1.0 to 3.5] | 1.13 [0.7 to 2.1] | 3.4 [1.85 to 5.45] | 3.4 [1.5 to 4.2]
  % T-lymphocytes that are T-helpers | 37.6 [26.6 to 48.9] | 41.4 [36.4 to 47.9] | 36.8 [33.6 to 44.2] | 39.8 [31.66 to 47.38] | 34.8 [29.1 to 41.0]
  % T-lymphocytes that are T-cytotoxic cells | 20.1 [16.0 to 28.8] | 24.8 [18.9 to 29.8] | 19.1 [15.2 to 23.4] | 22.46 [18.89 to 26.43] | 22.9 [20.1 to 27.7]
  % lymphocytes that are B-cells | 20.5 [13.6 to 31.6] | 17.3 [10.7 to 23.2] | 27.4 [21.3 to 33.0] | 14.18 [10.96 to 17.03] | 13.5 [10.3 to 17.4]
  % monocytes that are classical | 74.6 [67.0 to 81.4] | 81.2 [76.5 to 87.7] | 83.0 [75.7 to 85.7] | 78.0 [62.6 to 80.05] | 82.8 [78.8 to 88.1]
  % monocytes that are intermediate | 11.4 [7.17 to 18.5] | 7.02 [3.42 to 9.7] | 6.28 [4.93 to 12.4] | 12.6 [7.83 to 19.65] | 6.1 [4.2 to 9.5]
  % monocytes that are nonclassical | 2.03 [1.08 to 3.89] | 1.15 [0.56 to 2.43] | 2.16 [1.05 to 3.67] | 3.5 [1.39 to 5.3] | 1.1 [0.5 to 3.4]
  % neutrophils that express CD64 | 83.9 [74.0 to 93.7] | 5.55 [1.25 to 33.9] | 81.4 [44.7 to 94.3] | 0.35 [0.2 to 16.33] | 0.7 [0.3 to 1.6]
  % monocytes that express HLA-DR | 58.98 [28.76 to 96.64] | 88.54 [53.36 to 93.5] | 62.63 [44.07 to 95.6] | 86.4 [56.2 to 98.9] | 67.0 [56.3 to 97.1]
Statistical Analysis 1: Comparison: Patients With Sepsis, Day 1 vs Patients With Severe Bacterial Infection vs Patients With Severe Viral Infection; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Patients With Sepsis, Day 1 vs Patients With Severe Viral Infection vs Control Group; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Patients With Sepsis, Day 1 vs Patients With Sepsis, Day 7 vs Patients With Severe Bacterial Infection; Test type: Other; p < 0.02, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Patients With Sepsis on Day 1 | Patients With Sepsis on Day 7 | Patients With Severe Bacterial Infection | Patients With Severe Viral Infection | Control Group
All-Cause Mortality (participants affected / at risk) | 3/50 | 0/47 | 0/33 | 0/20 | 0/35
Serious Adverse Events (participants affected / at risk) | 3/50 | 0/47 | 0/33 | 0/20 | 0/35
Other Adverse Events (participants affected / at risk) | 0/50 | 0/47 | 0/33 | 0/20 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Sepsis on Day 1 (N=50) | Patients With Sepsis on Day 7 (N=47) | Patients With Severe Bacterial Infection (N=33) | Patients With Severe Viral Infection (N=20) | Control Group (N=35)
death (Infections and infestations) | 3 | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT05908162/Prot_SAP_000.pdf